CLINICAL TRIAL: NCT04423224
Title: Non-invasive Stroke Volume-based ﬂuid Management in Elderly Patients Undergoing Hip Fracture Surgery Under Spinal Anaesthesia
Acronym: AttikonHSV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Associate Professor of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AttikonHSV
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Fluid Management; Haemodynamic Instability

STUDY DESIGN:
Intervention Model Description: Control group Management of the hemodynamic status in the control group versus a goal directed group based on stroke volume variation protocol (with Nexfin monitor) in patients undergoing hip fracture fixation under spinal anesthesia
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group Management of the hemodynamic status in the control group will be performed in the discretion of the attending anesthesiologist, with the aim of keeping mean arterial pressure (MAP) > 65mmHg. The type and amount of delivered fluids, and vasoactive or inotropic drugs will be recorded.
  Interventions: Other: USUAL CARE - CONTROL
- GDFM (Active Comparator): Goal-directed fluid management group (GDFM). . Baseline SV will be measured after the patients will be turned to left/right position & before implementation of regional anesthesia. Fluid challenges of 250 ml will be repeated until SV fails to increase by 10%. At this point, preload is considered optimized and SV optimum is defined. SV trigger is defined as SV opt - 10%. N/S 250ml boluses will be administered when SV is below SV trigger. Inotropic drugs will be administered (dobutamine infusion at 0.2-10mcg/kg/min) if CO is below 3.5 L/min and vasopressors (phenylephrine bolus doses of 50-100mcg) if SV and CO are within the target range but MAP is below 65mmHg. Patients will be reassessed during the intraoperative period every 10 minutes . Except from the fluid boluses, all patients will be administered Ringer's lactate solution at an infusion rate of 2ml/kg/h.
  Interventions: Other: GDFM

INTERVENTIONS:
Other: GDFM — Stroke volume variation fluid management
  Arms: GDFM
Other: USUAL CARE - CONTROL — Usual care fluid management
  Arms: Control group

SUMMARY:
The study is going to be a single-centre prospective randomized trial. Patients will be randomly allocated to either control group (anesthetist-directed fluid therapy) or goal directed fluid therapy group, in which fluid therapy was guided by stoke volume (SV) algorithm with the use of Nexfin monitor. Primary outcome measures were the time to hospital discharge since surgery and the occurence of complications developed during the postoperative period. Secondary outcomes included the incidence of intraoperative hypotensive episodes (with MAP<65mmHg) in both groups and the requirement of vasoactive drugs to support blood pressure

DETAILED DESCRIPTION:
The study is going to be a single-centre prospective randomized trial in elderly patients undergoing hip fracture surgery under spinal anesthesia.

Patients will be randomly allocated to either control group (anesthetist-directed fluid therapy) or goal directed fluid therapy group, in which fluid therapy was guided by stoke volume (SV) algorithm with the use of Nexfin monitor.

In patients of the control group management of the hemodynamic status will be performed in the discretion of the attending anesthesiologist, with the aim of keeping mean arterial pressure (MAP) > 65mmHg. The type and amount of delivered fluids, and vasoactive or inotropic drugs will be recorded.

In Goal Directed Fluid Therapy group, fluid management will be guided by the Nexfin monitor, based on stroke volume of the patient under continuous tracking. Baseline SV will be measured after the patients will be turned to left/right position (at which they are going to stay throughout the whole procedure) and before the implementation of regional anesthesia. Fluid challenges of 250 ml will be repeated until the SV fails to increase by 10%. At this point, preload is considered optimized and SV optimum iss defined. SV trigger is defined as SV opt - 10%. After obtaining these values, the anesthetic and surgical interventions could proceed. During surgery, N/S 250ml boluses will be administered when SV is below SV trigger. Inotropic drugs will be administered (dobutamine infusion at 0.2-10mcg/kg/min) if CO is below 3.5 L/min and vasopressors (phenylephrine bolus doses of 50-100mcg) if SV and CO are within the target range but MAP is below 65mmHg.

Primary outcome measures were the time to hospital discharge since surgery and the occurence of complications developed during the postoperative period. Secondary outcomes included the incidence of intraoperative hypotensive episodes (with MAP<65mmHg) in both groups and the requirement of vasoactive drugs to support blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip fracture repair
* over 60 years of age
* American Society of Anesthesiologists (ASA) physical status II, III, IV

Exclusion Criteria:

* refusal or inability to consent,
* a plan for general anesthesia
* expected unreliable measurements of nexfin monitor (e.g. peripheral vascular disease, finger edema).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
days of hospitalization after surgery | 30 days
  days of hospitalization after the operation
complications | 30 days
  incidence of complications

SECONDARY OUTCOMES:
hypotension | during surgery
  incidence of hypotensive episodes (MAP < 65mmHg)
use of vasoactive agents | during surgery
  use of vasoactive agents (phenylephrine, dopamine) exact dose

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - 2nd Department of Anaesthesiology, Attikon Hospital, 1 Rimini str., Athens, Attica
  - 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens

IPD SHARING:
Plan to Share IPD: Undecided